CLINICAL TRIAL: NCT05095103
Title: Comparison of Lymphocyte Subset, Cytokine and Complement Profiles in Myasthenia Gravis of Different Severity, Disease Time-points, and Treatment History
Brief Title: Immune Profiles in Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other); Walton Centre NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); University College London Hospitals (Other); University Hospital Birmingham NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); King's College Hospital NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Cardiff University (Other)
Responsible Party: Principal Investigator, Katherine Dodd, Neurology Clinical Research Fellow and PhD Student, University of Manchester
Other Study IDs: NHS001843
Record Dates: First submitted 2021-09-28; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stable Immunosuppressed: Acetylcholine repector antibody positvie myasthenia gravis, stable for two years on prednsiolone <5mg/day and azathioprine or mycophenolate.
- Stable Non-immunosuppressed: Acetylcholine repector antibody positvie myasthenia gravis, stable for two years on ≤120mg pyridostigmine/day and no immunosuppression.
- Refractory: Acetylcholine repector antibody positvie myasthenia gravis, meeting the NHS England criteria for Rituximab
- Healthy Controls: No autoimmune disease or current solid organ or haematological malignancy.

SUMMARY:
The investigators aim to better describe the immune profile in myasthenia gravis (MG), including lymphocyte subset, cytokine and complement profiles; how they differ between patients of different severity, at times of disease exacerbation, and with different immunosuppressive treatments. The investigators hope to build a clearer picture of how different immune measures vary in MG, contributing to the understanding of the patho[physiology of the disease, and working towards a biomarker that might help clinicians optimise an individual's treatment.

the investigators aim to take into account the heterogeneity of MG by taking into account age of onset of MG (early vs late onset) and focussing on acetylcholine receptor antibody (AChR) positive, non-thymomatous MG aged 18-80.

DETAILED DESCRIPTION:
This study is designed to confirm and refine the knowledge around these changes in the immune profile, including lymphocyte subsets, and complement analysis, between different subgroups of patients with MG of different severity, different levels of immunosuppressive treatment, and at different time points in the disease course, ensuring these are put into the context of the patient's disease subtype (late-onset (LOMG) vs early-onset (EOMG)). This should enable us to understand more about the underlying immune changes in MG, how they relate to disease activity or severity, how this is impacted upon by immunosuppression, and guide us towards a markers for disease severity and effective immunosuppression that could be used in clinical practice, and help guide treatment decisions. One of the challenges in studying patients with MG with the relatively low prevalence of the condition, meaning it can be difficult to recruit large enough numbers of patients; the investigators will work with other tertiary neurology centres throughout England in order to meet recruitment targets.

The research project will consist of three work streams:

1. A one-off observational comparison of the immune profile of patients with different MG severity and in comparison to healthy controls.
2. A prospective observational study examining changes in lymphocyte subset, cytokine and complement profiles associated with clinical exacerbation of myasthenia gravis.
3. A prospective cohort study comparing lymphocyte subset, cytokine and complement profile with disease activity following B cell depletion for refractory myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

* All participants:
* Are able to give valid written consent
* are aged between the ages of 18 and 80

Stable Immunosuppressed

* Have a diagnosis of AChR positive myasthenia gravis (can be ocular, bulbar or generalised)
* MGFA Post-intervention Status MM or better with no clinical relapse for 2 years
* On either azathioprine or MMF along with ≤5mg/day of prednisolone
* No prednisolone dose increase or decrease in past 12 months
* No increase in azathioprine or MMF dose for 2 years (allowing for cessation for up to 1 month)

Stable Non-Immunosuppressed

* have a diagnosis of AChR positive myasthenia gravis (can be ocular, bulbar or generalised)
* MGFA Post-intervention Status MM or better on only low-dose cholinesterase inhibitors (≤<120 mg pyridostigmine/day) for over two years and ≤5mg/day of prednisolone for over two years.
* No prednisolone dose increase or decrease in past 12 months

Refractory

* have a diagnosis of AChR positive myasthenia gravis (can be ocular, bulbar or generalised)
* have been deemed eligible to be refractory to standard treatment and eligible for rituximab as per the NHS England criteria.

Exclusion Criteria for all participants:

* Are unable to give valid consent
* Co-existing autoimmune condition for which azathioprine or mycophenolate mofetil are treatments (e.g. inflammatory bowel disease, rheumatoid arthritis, neuromyotonia)
* Currently undergoing treatment for solid organ or haematological malignancy, or previous thymoma
* Clinical frailty scale ≥6

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acetylcholine receptor antibody positive myasthenia gravis
Sampling Method: Non-Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Primary outcome work stream 1 | Baseline
  Difference in CD19 count between cohorts
Primary outcome work stream 2 | Relapse within 18 months of recrutiment
  ● CD27 frequency (% of peripheral blood mononuclear cells) at clinical exacerbation of MG compared to when that patient was clinically stable.
Primary outcome work stream 3 | 12 months after B cell depletion
  ● CD27+ frequency (% of peripheral blood mononuclear cells) in MG patients who are symptomatic compared to those who are asymptomatic 12 months following B cell depletion.

SECONDARY OUTCOMES:
MG Composite Score | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups,
MGFA - Post Intervention status | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups
MG QOL-15r | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups
Acetylcholine receptor antibody titre | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups
Lymphocyte Count | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups
Number of relapses requiring hospital admission or rescue therapy | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups
Average daily dose of prednisolone over the three months prior to review | Baseline, at any clinical relapse within 18 months, 3,6 months after relapse in stable groups or 4 weeks, 6 and 12 months post rituximab in refractory groups

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Dodd, MBChB MRCP, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: No